CLINICAL TRIAL: NCT06567483
Title: A Comparison of Protein-bound and Large Molecular Weight Uremic Toxin Removals With Novel Super High-flux Dialyzer Between Hemodialysis and High Volume Online Hemodiafiltration Modalities : A Crossover Randomized Controlled Study
Brief Title: A Comparison of Protein-bound and Large Molecular Weight Uremic Toxin Removals With Novel Super High-flux Dialyzer Between Hemodialysis and High Volume Online HDF Modalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Rossanun Shoosanglertwijit, MD, Principle investigator, Chulalongkorn University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 051466
Record Dates: First submitted 2024-03-13; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Uremic; Toxemia
Keywords: Super High-flux dialyzers; Medium cut-off membrane; Protein bound uremic toxin; Indoxyl sulfate; Dialysate albumin loss; Albumin; Kappa free light chain; Lambda free light chain; Pre-dilution online HDF; Conventional hemodialysis
MeSH Terms: conditions — Toxemia

STUDY DESIGN:
Intervention Model Description: After a run-in period, the patients were randomly allocated to receive either 8-week of predilution hemodiafiltration using super-high flux, ELISIO-21HX, or hemodialysis using super-high flux as the control treatment. After a wash-out period of hemodiafiltration using high flux dialyzer, they were assigned to receive the other treatment for 8 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Predilution online hemodiafiltration (Experimental): The dialysis mode will be set as predilution online hemodiafiltration for 8 weeks.
  Interventions: Device: ELISIO21HX
- Hemodialysis (Active Comparator): The dialysis mode will be set as conventional hemodialysis for 8 weeks.
  Interventions: Device: ELISIO21HX

INTERVENTIONS:
Device: ELISIO21HX — Super-high flux dialyzers (ELISIO21HX) will be used. The blood flow rate and dialysate flow rate will be set as 400 and 800 ml/min respectively for 4 hours of dialysis.
  Other Names: Super-high flux dialyzer

SUMMARY:
The goal of this prospective, randomized, crossover study is to study about using super high-flux dialyzer in the chronic hemodialysis patients.

The main questions aim to answer are the reduction ratio of protein bound uremic toxins

Participants will undergone the pre-dilution online hemodiafiltration and conventional hemodialysis for each 8 weeks followed by washout phase for 4 weeks.

DETAILED DESCRIPTION:
Other secondary outcomes that the researcher wants to study are

1. The reduction ratio of Beta2microglobulin, kappa and lambda free light chain
2. Serum albumin and dialysate albumin loss
3. Quality of life, muscle mass and nutritional status of the patients

ELIGIBILITY:
Inclusion Criteria:

* Chronic hemodialysis patients in King Chulalongkorn Memorial hospital
* Residual renal function less than 100 ml/day

Exclusion Criteria:

* Dialyzer allergy
* Malnutrition requiring intradialytic parenteral nutrition
* Cirrhosis child C or decompensated cirrhosis
* Active uncontrolled infection
* Active cardiovascular disease
* Advanced stage malignancy
* Predicted to be undergone living related kidney transplant within 1 year

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Protein bound uremic toxin reduction ratio (percent) | 8 weeks
  The reduction ratio of indoxyl sulfate will be calculated as percent by pre and post dialysis data. The measurement will take place in the pre-dialysis of the first and the last time of intervention

SECONDARY OUTCOMES:
Beta2 microglobulin, kappa and lambda free light chain and urea reduction ratio (percent) | 8 weeks
  The reduction ratio of the beta2 microglobulin, kappa and lambda free light chain and urea will be measure at the first and the last time of intervention by pre and post dialysis level.
Serum albumin and dialysate albumin loss | 8 weeks
  Serum albumin will be followed at the midweek pre-dialysis at the first and 8th weeks of intervention.
  Dialysate albumin will also be assessed at the 1st and the 8th weeks.
Quality of life assessment in each group | 8 weeks
  Quality of life was assessed by the KDQOL36 questionnaire in each intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rossanun Shoosanglertwijit, Principal Investigator — Chulalongkorn University; Khajohn Tiranathanagul, Principal Investigator — Chulalongkorn University; Pajaree Chariyavilaskul, Principal Investigator — Chulalongkorn University
Locations (1):
- Faculty of Medicine Chulalongkorn university, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
Share only the results of the study.